CLINICAL TRIAL: NCT04222816
Title: Effect of Regulated Add -on Sodium Chloride Intake on Stabilization of Serum Lithium Concentration in Bipolar Disorder: A Randomized Controlled Trial
Brief Title: Effect of Regulated Add -on Sodium Chloride Intake on Stabilization of Serum Lithium Concentration in Bipolar Disorder
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: All India Institute of Medical Sciences, Bhubaneswar (Other)
Responsible Party: Principal Investigator, RITUPARNA MAITI, Additional Professor, All India Institute of Medical Sciences, Bhubaneswar
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IEC/AIIMS BBSR/PG Th/19-20/76
Record Dates: First submitted 2020-01-07; First posted 2020-01-10 (Actual); Last update posted 2022-01-25 (Actual); Status verified 2022-01

CONDITIONS: Bipolar Affective Disorder
Keywords: Bipolar affective disorder; Lithium; Manic depressive psychosis; Sodium chloride
MeSH Terms: conditions — Bipolar Disorder | interventions — Lithium Carbonate; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Randomized, open label, parallel group, active controlled clinical trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Lithium carbonate (Active Comparator): Lithium carbonate is prescribed 800-900 mg per day for 12 weeks.
  Interventions: Drug: Lithium Carbonate
- Add-on Sodium chloride (Experimental): Sodium chloride 1gm per day per will be prescribed along with Lithium carbonate 800-900 mg per day for 12 weeks.
  Interventions: Drug: Lithium Carbonate; Drug: Sodium chloride

INTERVENTIONS:
Drug: Lithium Carbonate — Lithium carbonate 800-900 mg orally daily for 12 weeks
Drug: Sodium chloride — Sodium chloride 1gm daily per orally for 12 weeks
  Arms: Add-on Sodium chloride

SUMMARY:
Bipolar affective disorder or manic -depressive psychosis (MDP) is a mood disorder affecting 2.4% of the global population . Lithium is considered as the "gold standard" for the treatment of bipolar disorder but the clinical use of lithium is often restricted due to its narrow therapeutic range and adverse effects.

In a published case report, Bleiwiss H found that sodium chloride supplementation diminished the adverse effects caused by lithium The literature search also revealed that till date, there is no published clinical study evaluating the effect of dietary intake of sodium in preventing the fluctuations of serum lithium level and lithium toxicity Therefore, a randomized clinical trial has been designed to evaluate the effect of regulated add -on dietary sodium chloride on serum lithium levels in bipolar disorder.

DETAILED DESCRIPTION:
Bipolar affective disorder or manic -depressive psychosis (MDP) is a mood disorder affecting 2.4% of the global population. Lithium is considered as the "gold standard" for the treatment of bipolar disorder but the clinical use of lithium is often restricted due to its narrow therapeutic range and adverse effects.One of the major adverse effects of lithium is nephrogenic diabetes insipidus which is due to long -term renal dysfunction.

In the initial months of lithium therapy, psychiatrists face difficulty in titrating the dose and stabilizing serum lithium level and this fluctuation of serum lithium level may be due to a lithium-induced sodium depleted state.

In a published case report, Bleiwiss H found that sodium chloride supplementation diminished the adverse effects caused by lithium. 8 In another case report, Tomita et al demonstrated that the change in sodium chloride intake can bring about changes in serum lithium and help in stabilizing the levels of serum lithium concentration.

As all the case reports are from abroad, the effect of dietary sodium on serum lithium level among Indian population is completely unknown. The literature search also revealed that till date, there is no published clinical study evaluating the effect of dietary intake of sodium in preventing the fluctuations of serum lithium level and lithium toxicity. Therefore, a randomized clinical trial has been designed to evaluate the effect of regulated add -on dietary sodium chloride on serum lithium levels in bipolar disorder. This study may help to explore the role of add -on sodium chloride in decreasing the fluctuations in the serum lithium level and improving the clinical outcome of patients with bipolar disorders.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 -60 years, of either sex with the clinical diagnosis of bipolar disorder (DSM V) who are on maintenance lithium therapy for ≥ 1month and ≤ 6 months.
* Patients with normal serum sodium level (135 -145 mEq/L) and serum lithium in the optimum therapeutic range (<0.6 mEq/ L or >0.8 mEq/ L) .

Exclusion Criteria:

* Patients with comorbidities like other psychiatric disorder s, organicity, substance abuse, personality disorder, intellectual disability and other neurotic disorders .
* Patients with any renal, cardiovascular, neurologica l, endocrinal and hepatic dysfunction.
* Patients suffering from diarrhoea, dehydration
* History of any invasive neurosurgical/ non -invasive neuropsychiatric procedure.
* Medication history of psychoactive or central nervous system depressant drugs.
* Patients who are on NSAIDs, ACE inhibitors, antiarrhythmics, diuretics and neuromuscular blocking agents .
* Pregnant and nursing women .
* Patients with drug/alcohol abuse.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2020-01-16 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-01-07 (Actual)

PRIMARY OUTCOMES:
Difference in percentage of bipolar patients showing fluctuation in serum lithium level | 12 weeks
  Serum lithium level will be done by electrolyte analyzer. The patients showing fluctuations ( fluctuation is defined as serum lithium <0.6 mEq/ L or >0.8 mEq/ L in maintenance phase) in serum lithium level between the groups over 12 weeks.

SECONDARY OUTCOMES:
Serum sodium | 12 weeks
  Will be done by electrolyte analyzer.
Serum Potassium | 12 weeks
  Will be done by electrolyte analyzer.
Serum creatinine | 12 weeks
  Will be done by autoanalyser.
Serum aldosterone | 12 weeks
  Will be done by commercially available ELISA kit.
ECG changes | 12 weeks
  ECG changes for lithium toxicity (T wave inversion, PR prolongation, QT prolongation), hyponatremia (P wave alterations), hypernatremia (short PR interval and diffuse ST depression) will be looked for
Serum Lithium | 12 weeks
  Will be done by electrolyte analyzer.

CONTACTS AND LOCATIONS:
Overall Officials: DEBASISH HOTA, DM, Study Director — PROFESSOR AND HEAD OF THE DEPARTMENT
Locations (1):
- Aiims Bhubaneswar, Khordha, Odisha, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Merikangas KR, Jin R, He JP, Kessler RC, Lee S, Sampson NA, Viana MC, Andrade LH, Hu C, Karam EG, Ladea M, Medina-Mora ME, Ono Y, Posada-Villa J, Sagar R, Wells JE, Zarkov Z. Prevalence and correlates of bipolar spectrum disorder in the world mental health survey initiative. Arch Gen Psychiatry. 2011 Mar;68(3):241-51. doi: 10.1001/archgenpsychiatry.2011.12. PMID 21383262
- [Background] Bleiweiss H. Salts supplements with lithium. Lancet. 1970 Feb 21;1(7643):416. doi: 10.1016/s0140-6736(70)91550-3. No abstract available. PMID 4189720
- [Background] Tomita T, Goto H, Sumiya K, Yoshida T, Tanaka K, Kohda Y. Stabilization of the Serum Lithium Concentration by Regulation of Sodium Chloride Intake: Case Report. Yakugaku Zasshi. 2016;136(3):517-21. doi: 10.1248/yakushi.15-00256. PMID 26935095
- [Background] Demers RG, Heninger GR. Sodium intake and lithium treatment in mania. Am J Psychiatry. 1971 Jul;128(1):100-4. doi: 10.1176/ajp.128.1.100. No abstract available. PMID 4949647
- [Background] Selvarajan S, Manohar H, Das S, Sakkarabani P, Kandasamy P. Lithium prophylaxis in early-onset Bipolar disorder: a descriptive study. Asian J Psychiatr. 2019 Aug;44:172-174. doi: 10.1016/j.ajp.2019.07.053. Epub 2019 Jul 30. PMID 31394485
- [Background] Tondo L, Vazquez GH, Baldessarini RJ. Depression and Mania in Bipolar Disorder. Curr Neuropharmacol. 2017 Apr;15(3):353-358. doi: 10.2174/1570159X14666160606210811. PMID 28503106
- [Background] Kessler RC, Ormel J, Petukhova M, McLaughlin KA, Green JG, Russo LJ, Stein DJ, Zaslavsky AM, Aguilar-Gaxiola S, Alonso J, Andrade L, Benjet C, de Girolamo G, de Graaf R, Demyttenaere K, Fayyad J, Haro JM, Hu Cy, Karam A, Lee S, Lepine JP, Matchsinger H, Mihaescu-Pintia C, Posada-Villa J, Sagar R, Ustun TB. Development of lifetime comorbidity in the World Health Organization world mental health surveys. Arch Gen Psychiatry. 2011 Jan;68(1):90-100. doi: 10.1001/archgenpsychiatry.2010.180. PMID 21199968
- [Background] Murthy RS. National Mental Health Survey of India 2015-2016. Indian J Psychiatry. 2017 Jan-Mar;59(1):21-26. doi: 10.4103/psychiatry.IndianJPsychiatry_102_17. No abstract available. PMID 28529357
- [Background] Mandal S, Mamidipalli SS, Mukherjee B, Hara SKH. Perspectives, attitude, and practice of lithium prescription among psychiatrists in India. Indian J Psychiatry. 2019 Sep-Oct;61(5):451-456. doi: 10.4103/psychiatry.IndianJPsychiatry_451_18. PMID 31579157
- [Derived] George S, Maiti R, Mishra BR, Jena M, Mohapatra D. Effect of regulated add-on sodium chloride intake on stabilization of serum lithium concentration in bipolar disorder: A randomized controlled trial. Bipolar Disord. 2023 Feb;25(1):66-75. doi: 10.1111/bdi.13276. Epub 2022 Nov 25. PMID 36409058